CLINICAL TRIAL: NCT05971693
Title: Safety and Effectiveness Evaluation of the OMNYPULSE Catheter With the TRUPULSE Generator for Treatment of Paroxysmal Atrial Fibrillation (PAF)
Brief Title: A Study For Treatment of Paroxysmal Atrial Fibrillation (PAF) With the OMNYPULSE Catheter and the TRUPULSE Generator
Acronym: Omny-IRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202201; BWI202201 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- OMNYPULSE Bi-Directional Catheter with TRUPULSE Generator (Experimental): Participants with symptomatic paroxysmal atrial fibrillation (PAF) will undergo the ablation procedure with OMNYPULSE bi-directional catheter used in combination with the TRUPULSE generator for pulmonary vein isolation (PVI).
  Interventions: Device: OMNYPULSE Bi-Directional Catheter with TRUPULSE Generator

INTERVENTIONS:
Device: OMNYPULSE Bi-Directional Catheter with TRUPULSE Generator — Participants will undergo catheter ablation with the PF ablation system consisting of the TRUPULSE generator (delivers PF energy through the study catheter) and the OMNYPULSE bi-directional catheter (indicated for use in catheter-based cardiac electrophysiological mapping [stimulating and recording] and, when used with a Generator, for cardiac ablation).

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the ablation system (OMNYPULSE Bi-directional catheter and TRUPULSE generator) when used for isolation of the atrial pulmonary veins (PVs) in treatment of participants with paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Symptomatic paroxysmal atrial fibrillation (PAF) defined as as atrial fibrillation (AF) that terminates spontaneously or with intervention within 7 days of onset. This PAF is considered to be symptomatic if symptoms related to AF are experienced by the participant
* Selected for AF ablation procedure by pulmonary vein isolation (PVI)
* Willing and capable of providing consent
* Able and willing to comply with all pre-, post- and follow-up testing and requirements

Exclusion Criteria:

* Previously known AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause (example, documented obstructive sleep apnea, acute alcohol toxicity, morbid obesity [body mass index greater than {>} 40 kilograms per meter square {kg/m^2}]), renal insufficiency (with an estimated creatinine clearance less than (<) 30 milliliters per minute per 1.73 meter square [mL/min/1.73 m^2])
* Previous left atrium (LA) ablation or surgery
* Participants known to require ablation outside the PV region (example, atrioventricular reentrant tachycardia, atrioventricular nodal re-entry tachycardia, atrial tachycardia, ventricular tachycardia and Wolff-Parkinson-White)
* Previously diagnosed with persistent AF (> 7 days in duration)
* Severe dilatation of the left atrium (LA) (left anterior descending artery [LAD] >50 millimeter [mm] antero-posterior diameter in case of transthoracic echocardiography [TTE])
* Presence of LA thrombus
* Severely compromised left ventricular ejection fraction (left ventricular ejection fraction [LVEF] <40 percentage [%])
* Uncontrolled heart failure or New York Heart Association (NYHA) Class III or IV
* History of blood clotting, bleeding abnormalities or contraindication to anticoagulation (heparin, warfarin, or dabigatran)
* History of a documented thromboembolic event (including transient ischemic attack [TIA]) within the past 6 months
* Previous percutaneous coronary intervention (PCI) / myocardial infarction (MI) within the past 2 months
* Previous coronary artery bypass grafting (CABG) in conjunction with valvular surgery, cardiac surgery (example, ventriculotomy, atriotomy) or valvular cardiac (surgical or percutaneous) procedure
* Unstable angina pectoris within the past 6 months
* Anticipated cardiac transplantation, cardiac surgery, or other major surgery within the next 12 months
* Significant pulmonary disease (example, restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
* Known significant pulmonary vein (PV) anomaly that in the opinion of the investigator would preclude enrollment in this study
* Prior diagnosis of pulmonary vein stenosis
* Pre-existing hemi diaphragmatic paralysis
* Acute illness, active systemic infection, or sepsis
* Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation
* Severe mitral regurgitation
* Presence of implanted pacemaker or implantable cardioverter-defibrillator (ICD) or other implanted metal cardiac device that may interfere with the pulsed electric field energy
* Presence of a condition that precludes vascular access (such as Inferior Vena Cava [IVC] filter)
* Significant congenital anomaly or a medical problem that in the opinion of the investigator would preclude enrollment in this study
* Categorized as vulnerable population and requires special treatment with respect to safeguards of well-being
* Current enrollment in an investigational study evaluating another device or drug
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of child-bearing age and plan on becoming pregnant during the course of the clinical investigation
* Life expectancy less than 12 months
* Presenting contra-indications for the devices used in the study, as indicated in the respective Instructions For Use (IFU)
* Known contraindication for magnetic resonance imaging (MRI) such as use of contrast agents due to advanced renal disease, claustrophobia etcetra. (at principle investigator [PI] discretion)
* Presence of iron-containing metal fragments in the body
* Known unresolved pre-existing neurological deficit
* Known uncontrolled significant gastroesophageal reflux disease (GERD)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Primary Adverse Events (PAE's) | 7 days post-ablation procedure on Day 0 (up to Day 7)
  Number of Participants with incidence of PAEs (within 7 days following the ablation procedure) will be reported. PAE's will include the following adverse events atrio-esophageal fistula, phrenic nerve paralysis, cardiac tamponade/perforation, pulmonary vein stenosis, device or procedure related death, stroke/cerebrovascular accident (CVA), major vascular access complication/bleeding, thromboembolism, myocardial infarction, transient ischemic attack (TIA), pericarditis, heart block, pulmonary edema (respiratory insufficiency) and vagal nerve injury/gastroparesis.
Percentage of Participants with Acute Effectiveness | Immediate post-procedure
  Percentage of participants with acute effectiveness will be reported. Acute effectiveness is an electrical isolation of clinically relevant targeted pulmonary veins (PVs) (confirmed by entrance block) after adenosine/isoproterenol challenge at the end of the index ablation procedure. Use of a non-study device to achieve PV isolation is considered an acute procedural failure.

SECONDARY OUTCOMES:
12-month Effectiveness: Number of Participants who Achieved Freedom from Documented Atrial Arrhythmia Episodes During the Effectiveness Evaluation period (AF, AT or AFL of Unknown Origin) within Day 91 to Day 365 Post Index Procedure | Within Day 91 to Day 365 post-ablation procedure (on Day 1)
  12-month effectiveness: Number of participants rate of Freedom from documented (symptomatic and asymptomatic) Atrial Arrhythmia (Atrial Fibrillation [AF], Atrial Tachycardia [AT] or Atrial Flutter [AFL] of unknown origin) episodes assessed during the effectiveness evaluation period (Day 91 to Day 365 days post index procedure will be reported. Freedom from atrial arrhythmia will be reported based on electrocardiographic data (greater than or equal to [>=30] seconds on arrhythmia monitoring device) during the effectiveness evaluation period on or off antiarrhythmic therapy. Acute procedural failure (that is, failure to achieve entrance block with the study device in any of the clinically relevant targeted PVs) will also be deemed a 12- month effectiveness failure.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc., a division of Johnson & Johnson Clinical Trial, Study Director — Biosense Webster, Inc., a division of Johnson & Johnson
Locations (13):
- Belgium (4):
  - AZORG campus Aalst Moorselbaan, Aalst
  - AZ Sint-Jan, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- KBC Split, Split, Croatia
- Czechia (2):
  - IKEM, Prague
  - Nemocnice na Homolce, Prague
- MVZ CCB Frankfurt und Main Taunus GbR, Frankfurt a.M., Germany
- Generale Regionale F. Miulli, Acquaviva delle Fonti, Italy
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Duytschaever M, Grimaldi M, De Potter T, Verma A, Macle L, Kautzner J, Linz D, Anic A, Van Herendael H, Rackauskas G, Neuzil P, Chun J, Schmidt B, Knecht S, Almorad A, Berte B, Reddy VY, Vijgen J. PVI With CF-Sensing Large-Tip Focal PFA Catheter With 3D Mapping for Paroxysmal AF: Omny-IRE 3-Month Results. JACC Clin Electrophysiol. 2025 Aug;11(8):1769-1782. doi: 10.1016/j.jacep.2025.04.008. Epub 2025 Apr 25. PMID 40340298